CLINICAL TRIAL: NCT06233994
Title: A Study Evaluating the Efficacy and Safety of ZG005 in Combination With Donafenib Tosilate Tablets or Bevacizumab as First-line Treatment in Patients With Advanced Hepatocellular Carcinoma
Brief Title: A Study Evaluating the Efficacy and Safety of ZG005 in Combination With Donafenib or Bevacizumab in Patients With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changsha Taihe Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZG005-IIT-001
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — Injections; donafenib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZG005+Donafenib (Experimental): Participants will receive ZG005 plus Donafenib until unacceptable toxicity or loss of clinical benefit.
  Interventions: Biological: ZG005 Powder for Injection; Drug: Donafenib Tosilate Tablets
- ZG005+Bevacizumab (Experimental): Participants will receive ZG005 plus bevacizumab until unacceptable toxicity or loss of clinical benefit.
  Interventions: Biological: ZG005 Powder for Injection; Biological: Bevacizumab

INTERVENTIONS:
Biological: ZG005 Powder for Injection — ZG005 will be administered at a dose of 10 mg/kg by intravenous (IV) infusion, once every 3 weeks (Q3W).
  Other Names: ZG005
Drug: Donafenib Tosilate Tablets — Donafenib will be administered at a dose of 0.2 g by orally, Bis in die(Bid).
  Other Names: Donafenib
  Arms: ZG005+Donafenib
Biological: Bevacizumab — Bevacizumab will be administered at a dose of 15 mg/kg by IV infusion, once every 3 weeks (Q3W).
  Arms: ZG005+Bevacizumab

SUMMARY:
This is a randomized, open-label study to evaluate the safety and efficacy of ZG005 in combination with Donafenib or Bevacizumab in patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age.
* Fully understand the study and voluntarily sign the informed consent form.
* Histologically or cytologically confirmed diagnosis of metastatic or unresectable hepatocellular carcinoma (HCC).
* Life expectancy >= 3 months.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

Exclusion Criteria:

* Fibrolamellar or sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Patients were deemed unsuitable for participating in the studyl by the investigator for any reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to approximately 2 years
  The sum of the proportions of subjects who achieved CR or PR in imaging evaluation as assessed by the investigator based on RECIST1.1 criteria.
Progression Free Survival (PFS) | up to approximately 2 years
  Time from first dose of the investigational drug to PD or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Chai, Principal Investigator — Changsha Taihe Hospital
Locations (1):
- Changsha Taihe Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No